CLINICAL TRIAL: NCT01095237
Title: Multicenter, Clinical Pilot-Study of ProEndoTecc Vascular Grafts (6, 7 or 8 mm Diameter) as Superficial Femoral Artery Bypass/Interponate
Brief Title: Clinical Pilot-Study of ProEndoTecc Vascular Grafts as Superficial Femoral Artery Bypass / Interponate
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study has been halted due to safety reasons
Sponsor: NonWoTecc Medical GmbH (Industry)
Collaborators: MDT Medical Device Testing GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: mdt-09k006
Record Dates: First submitted 2010-03-23; First posted 2010-03-30 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Peripheral Arterial Disease; Peripheral Vascular Disease
Keywords: Peripheral Arterial Disease; Peripheral Vascular Disease; PAD; vascular prosthesis; revascularization; patency; blood vessel; Rutherford; ABI; Ankle Brachial Index; Vascular Graft; Carbothane; ProEndoTecc; implantation
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: ProEndoTecc Vascular Graft — Implantation of the device as an interponate / bypass of the superficial femoral artery
  Other Names: ProEndoTecc Vascular Graft Prosthesis

SUMMARY:
This is a multi-center, clinical pilot-study of ProEndoTecc Vascular Grafts (6, 7 or 8 mm Diameter) as superficial femoral artery bypass/interponate.

The aim of this study is to demonstrate safety of implantation, patency and durability of a new type of vascular graft.

ELIGIBILITY:
Inclusion Criteria:

* Female or male patient from 18 to 89 years of age
* Superficial femoral artery occlusion from 5 to 40 cm in length (above the knee joint),
* Patient must present with intermittent claudication, with resistance to medical therapy and exercise or critical ischemia,
* Patient has Rutherford grade 3, 4, or 5 occlusive vascular disease,
* Women of childbearing age must have negative pregnancy test prior to inclusion

Exclusion Criteria:

* Bleeding diathesis
* Patient has known coagulation disorders including hypercoagulability
* Presence of one or several previously placed endo-prosthesis or grafts in the diseased extremity (below iliacs)
* Other than 6-8 mm diameter graft is needed.
* Patients PAD state is in Fontaine Grade IV, Rutherford Grade 6 (Patient has active infection or pronounced necrosis in the region of graft placement)
* Patient has an acute embolic arterial occlusion
* Life-expectancy less than 6 month due to co-morbidity or other situation that would make the patient an unlikely candidate for follow-up visits
* Patient had percutaneous transluminal angioplasty at the implant site within the previous 30 days
* Participation in another clinical study less than 30 days prior to inclusion
* Patient is in need of, or is scheduled for, a cardiac surgical procedure or a different vascular surgical procedure
* Pregnant or breast feeding female patients
* Multiple graft (implant) needed
* Patients unable to understand the full meaning of the informed consent
* Subjects who, in the opinion of the investigator, will be inappropriate for inclusion into this trial or will not comply with requirements of the study
* Subjects who are imprisoned (according to MPG §20.3)
* Patients who are lawfully kept in an institution
* Participation in this trial at an earlier stage
* Current participation in another clinical trial

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Primary patency of device | 6, 12, 24 months after implatation
  Primary Patency of treated arterial segment at 6 month after intervention. Primary Patency is defined by objective demonstration via colour-coded Doppler sonography or angiography that the entire length of the graft remain patent with no further intervention required for symptomatic recurrent disease.
  In case this information is not available, primary patency might be declared, if any the following criteria are fulfilled: Present ABI increased of ≥0.1 compared to preoperative status Present PAD-Grade according to Rutherford increased by one degree Palpable pulse distal of prosthesis.

SECONDARY OUTCOMES:
Guarding Safety variables | 6,12, 24 months after implantation
  * Peri-interventional monitoring resp. haemorrhages, haematomas
  * Aneurysm in the grafted segment
  * Fistula to the grafted segment
  * Fibrosis at and around implantation site
  * Death

CONTACTS AND LOCATIONS:
Locations (12):
- Germany (12):
  - Staedtisches Klinikum Karlsruhe gGmbH, Karlsruhe, Baden-Wurttemberg
  - Klinikum Deggendorf, Dpt. of Vascular- and Endovascular Surgery, Deggendorf, Bavaria
  - Hospital Muenchen-Pasing, Munich, Bavaria
  - Klinikum Nuernberg Sued Dpt. of Vascular Surgery, Nuremberg, Bavaria
  - Krankenhaus Barmherzige Brüder, Dpt. of Vascular Surgery, Regensburg, Bavaria
  - Klinik fuer Gefaesschirurgie St-Bonifatius-Hospital Lingen, Lingen, Lower Saxony
  - Luisenhospital Dpt. of Vascular Surgery, Aachen, North Rhine-Westphalia
  - Gefaesschirurgische Klinik St-Marienhospital Bonn, Bonn, North Rhine-Westphalia
  - Knappschaftskrankenhaus Bottrop Dpt. of Vascular Surgery, Bottrop, North Rhine-Westphalia
  - Clinic and Polyclinic for Vascular Surgery, Cologne, North Rhine-Westphalia
  - Evangelisches Krankenhaus Dpt. of Vascular Surgery, Mülheim, North Rhine-Westphalia
  - Sana Clinic Remscheid Dpt. of Vascular Surgery, Remscheid, North Rhine-Westphalia